CLINICAL TRIAL: NCT04725084
Title: Comparison of Non-invasive Oxygenation Strategies in ICU Patients Admitted for Covid-19 Acute Respiratory Distress Syndrome
Brief Title: Comparison of Non-invasive Oxygenation Strategies in Patients Admitted for Covid-19 Acute Respiratory Distress Syndrome
Acronym: SONIC-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-CHITS-001
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-10

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Keywords: Novel coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Acute respiratory distress syndrome; High flow nasal canula oxygen; Non-invasive ventilation; Continuous positive airway pressure
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High Flow Nasal Cannula oxygen therapy treatment: Patients treated only by high flow nasal cannula oxygen therapy
  Interventions: Other: Use of High Flow Nasal Cannula alone
- Non-Invasive Ventilation treatment: Patients treated by non-invasive ventilation (combined or not with HFNC)
  Interventions: Other: Use of Non-invasive Ventilation
- Continuous Positive Airway Pressure treatment: Patients treated by continuous positive airway pressure (combined or not with HFNC)
  Interventions: Other: Use of Continuous Positive Airway Pressure

INTERVENTIONS:
Other: Use of High Flow Nasal Cannula alone — Use of high flow nasal cannula oxygen therapy alone
  Groups: High Flow Nasal Cannula oxygen therapy treatment
Other: Use of Non-invasive Ventilation — Use of non-invasive ventilation combined or not with high flow nasal cannula oxygen therapy
  Groups: Non-Invasive Ventilation treatment
Other: Use of Continuous Positive Airway Pressure — Use of continuous positive airway pressure combined or not with high flow nasal cannula oxygen therapy
  Groups: Continuous Positive Airway Pressure treatment

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is the main clinical presentation of SARS-CoV-2 (Covid-19) infected patients admitted in Intensive Care Unit (ICU).

During the first phase of the outbreak (between February and May 2020), the use of invasive Mechanical Ventilation (MV) was largely required with 63% of ICU patients intubated in the first 24 hours after admission and up to 80% of patients during the overall ICU stay. Mortality was especially higher when using MV in the first 24 hours. In contrast, the use of non-invasive oxygenation strategies in the first 24 hours was only 19% for High Flow Nasal Cannula oxygen therapy (HFNC) and 6% for Non-Invasive Ventilation (NIV).

Several non-invasive oxygenation strategies were proposed in order to delay or avoid MV in ICU patients suffering from Covid-19 ARDS. The use of HFNC became the recommended oxygenation strategy, based in particular on publications prior to the outbreak. The use of NIV or Continuous Positive Airway Pressure (CPAP) combined with HFNC have also been proposed. Although these non-invasive oxygenation strategies seem widely used in the second phase of the outbreak, they have not yet confirmed their clinical impact on MV requirement and patient's outcome. Moreover, no comparison has been made between these different non-invasive oxygenation strategies.

The aim of this study is to compare different non-invasive oxygenation strategies (HFNC, NIV, CPAP) on MV requirement and outcome in ICU patients treated for ARDS related to Covid-19.

DETAILED DESCRIPTION:
Retrospective multicenter observational registry in French intensive care unit including all consecutive patients admitted for acute respiratory distress syndrome related to SARS-CoV-2 pneumonia between1st July and 31th December 2020.

Patients characteristics, ICU treatments and outcome will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted in intensive care unit because of a SARS-CoV-2 infection confirmed by PCR wherever was collected the analyzed sample
* acute respiratory distress syndrome according to Berlin criteria
* age superior or equal to 18 years old

Exclusion Criteria:

* patient opposition to participate in the study
* patients under judicial protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted in intensive care unit for an acute respiratory distress syndrome related to a documented SARS-CoV-2 disease
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Refractory hypoxemia | Through Intensive Care Unit stay, an average of 15 days
  Rate of refractory hypoxemia outcome defined by invasive Mechanical Ventilation (endotracheal intubation) requirement or death of non-intubated patients because of therapeutical limitation

SECONDARY OUTCOMES:
Mechanical Ventilation free days | Through Intensive Care Unit stay, up to 1 month
  Numbers of days without invasive mechanical ventilation during ICU stay and until ICU discharge
Survival at ICU discharge | At the moment of Intensive care unit discharge, up to 1 month
  Rate of patients alive at the moment of intensive care unit discharge
ICU length of stay | At the moment of Intensive care unit discharge, up to 1 month
  Number of days spent in Intensive care unit
Complications during ICU stay | Through Intensive Care Unit stay, up to 1 month
  Number of complications during intensive care unit stay: pneumothorax, pneumomediastinum
Delay between admission and intubation | Through Intensive Care Unit stay, up to 1 month
  Period of time (in hours or days) between admission in Intensive Care Unit and intubation requirement with invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chelly, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (4):
- France (4):
  - Centre Hospitalier de Bethune, Béthune, Hauts-de-France
  - Grand Hôpital de l'Est Francilien, Jossigny, Seine-et-Marne
  - Groupe Hospitalier Sud Ile de France, Melun, Seine-et-Marne
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] COVID-ICU Group on behalf of the REVA Network and the COVID-ICU Investigators. Clinical characteristics and day-90 outcomes of 4244 critically ill adults with COVID-19: a prospective cohort study. Intensive Care Med. 2021 Jan;47(1):60-73. doi: 10.1007/s00134-020-06294-x. Epub 2020 Oct 29. PMID 33211135
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Background] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Background] Nightingale R, Nwosu N, Kutubudin F, Fletcher T, Lewis J, Frost F, Haigh K, Robinson R, Kumar A, Jones G, Brown D, Abouyannis M, Beadsworth M, Hampshire P, Aston S, Gautam M, Burhan H. Is continuous positive airway pressure (CPAP) a new standard of care for type 1 respiratory failure in COVID-19 patients? A retrospective observational study of a dedicated COVID-19 CPAP service. BMJ Open Respir Res. 2020 Jul;7(1):e000639. doi: 10.1136/bmjresp-2020-000639. PMID 32624495
- [Background] Avdeev SN, Yaroshetskiy AI, Tsareva NA, Merzhoeva ZM, Trushenko NV, Nekludova GV, Chikina SY. Noninvasive ventilation for acute hypoxemic respiratory failure in patients with COVID-19. Am J Emerg Med. 2021 Jan;39:154-157. doi: 10.1016/j.ajem.2020.09.075. Epub 2020 Oct 1. PMID 33067061
- [Result] Chelly J, Coupry LM, van Phach Vong L, Kamel T, Marzouk M, Terzi N, Bruel C, Autret A, Garnero A, Arnal JM. Comparison of high-flow nasal therapy, noninvasive ventilation, and continuous positive airway pressure on outcomes in critically ill patients admitted for COVID-19 with acute respiratory failure. Minerva Anestesiol. 2023 Jan-Feb;89(1-2):66-73. doi: 10.23736/S0375-9393.22.16918-X. Epub 2022 Nov 30. PMID 36448989